CLINICAL TRIAL: NCT00542594
Title: A Report Upon a Cohort of Post-menopausal Women Followed up After Treatment With Anastrozole as Adjuvant Therapy for Hormone-dependant Breast Cancer. Long-term Tolerance Evaluation
Brief Title: Survey in Post-menopausal Women Followed up After Treatment With Anastrozole as Adjuvant Therapy
Acronym: ARIES
Status: Terminated | Type: Observational
Why Stopped: No results are avaialble as the study did not complete according to the protocol
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OFR-ARI-2005/1
Record Dates: First submitted 2007-10-09; First posted 2007-10-11 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; anastrozole
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this survey is to describe long-term tolerance as seen under current conditions of use for anastrozole.

ELIGIBILITY:
Inclusion Criteria:

* woman treated with anastrozole as adjuvant therapy for hormone-dependant breast cancer in post-menopausal women with positive hormone-receptors

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Woman seen by their physician in the current care setting and for whom a treatment with anastrozole is decided by the physician (adjuvant treatment of breast cancer in postmenopausal women with hormone receptor positive status)
Sampling Method: Probability Sample
Enrollment: 1840 (Actual)
Dates: Start 2005-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca France Medical Director, Study Director — AstraZeneca